CLINICAL TRIAL: NCT00146016
Title: Study on Chronic Hepatitis C Treatment With Interferon Alpha, Ribavirin and Amantadine in Naive Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIRA-study
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2005-09-05 (Estimated); Status verified 2005-09

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic Hepatitis C; Amantadine; Triple therapy
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Amantadine

INTERVENTIONS:
Drug: Amantadine

SUMMARY:
* Adding Amantadine to standard anti-viral treatment can improve sustained response rates in patients with chronic hepatitis C

DETAILED DESCRIPTION:
The CIRA-study is a double blind, placebo controlled, randomised, multicentre study in previously untreated patients suffering from chronic hepatitis C comparing double therapy, consisting of (PEG-)interferon alpha 2b ((PEG)Intron-A®) and ribavirin (Rebetol®), with triple therapy, consisting of (PEG-)interferon alpha 2b, ribavirin and amantadine, for 52 weeks. Follow-up is completed at week 104. 150 Subjects per treatment group will be included. Patients will be stratified before randomisation according to genotype (1 versus non-1). Viral load will not be a discriminating factor.

The aim is to investigate the efficacy of the adjunct amantadine to the currently used combination therapy with interferon alpha and ribavirin.

ELIGIBILITY:
Inclusion Criteria:

* Anti-HCV positivity >6 months
* ALT and/or AST elevation on at least once in the previous 6 months
* Positive HCV-RNA
* Liver biopsy within one year before the start of therapy in non- cirrhosis. In the case of known cirrhosis, liver biopsy is not necessary
* Intention to be treated and participate treatment
* Obtained written informed consent

Exclusion Criteria:

* Age < 18 years
* Pregnancy or intention to get pregnant within the 12 months period of treatment and up to 6 months after discontinuation of therapy, no adequate contraception, lactation
* Men not practicing or willing to practice acceptable methods of contraception during the treatment period and up to 6 months after discontinuation of therapy
* Life expectancy < 1 year
* Child Pugh B or C (Appendix III)
* Creatinine > 150 μmol/L or > 1.70 mg/dl
* Haemoglobulin < 6.5 mmol/l or < 10.5 g/dl
* White blood cell count < 2,5 x 109/L, neutrophil < 1,5 x 109/L
* Platelet count < 70 x 109/L
* HIV positivity
* Chemotherapy, systematical antiviral treatment during the 6 months prior to study entry
* Other serious disease (e.g. malignancy, uncontrolled myocardial disease or severe arrhythmias)
* Active uncontrolled psychiatric disorders and suicidal leanings
* Patients with a history of uncontrolled seizure or other significant CNS dysfunction
* Any condition which in the opinion of the (co-)investigator might interfere with the evaluation of the study objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390
Dates: Start 2000-02; Study Completion 2007-01

PRIMARY OUTCOMES:
Response rate at end of treatment and end of follow-up (sustained response rate)

CONTACTS AND LOCATIONS:
Overall Officials: Karel v. Erpecum, MD, PhD, Principal Investigator — UMC Utrecht, dept. Gastroenterology; Melvin Samsom, MD, PhD, Principal Investigator — UMC Utrecht, dept gastroenterology
Locations (1):
- UMC Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Background] Berg T, Kronenberger B, Hinrichsen H, Gerlach T, Buggisch P, Herrmann E, Spengler U, Goeser T, Nasser S, Wursthorn K, Pape GR, Hopf U, Zeuzem S. Triple therapy with amantadine in treatment-naive patients with chronic hepatitis C: a placebo-controlled trial. Hepatology. 2003 Jun;37(6):1359-67. doi: 10.1053/jhep.2003.50219. PMID 12774015
- [Background] Brillanti S, Levantesi F, Masi L, Foli M, Bolondi L. Triple antiviral therapy as a new option for patients with interferon nonresponsive chronic hepatitis C. Hepatology. 2000 Sep;32(3):630-4. doi: 10.1053/jhep.2000.16235. PMID 10960460
- [Background] Younossi ZM, McCullough AC, Barnes DS, Post A, Ong JP, O'Shea R, Martin LM, Bringman D, Farmer D, Levinthal G, Mullen KD, Carey WD, Tavill AS, Ferguson R, Gramlich T. Pegylated interferon alpha-2b, ribavirin and amantadine for chronic hepatitis C. Dig Dis Sci. 2005 May;50(5):970-5. doi: 10.1007/s10620-005-2673-y. PMID 15906777
- [Derived] Van Vlerken LG, Van Soest H, Janssen MP, Boland GJ, Drenth JP, Burger DM, Siersema PD, Van Erpecum KJ. Suboptimal endogenous erythropoietin response in chronic hepatitis C patients during ribavirin and PEG interferon treatment. Eur J Gastroenterol Hepatol. 2010 Nov;22(11):1308-15. doi: 10.1097/MEG.0b013e32833e784d. PMID 20729740